CLINICAL TRIAL: NCT01768884
Title: Phase IIa Prospective, Double Blind, Randomized Single-Center, Evaluation of the Safety and Tolerability of Nitric Oxide Given Intermittently Via Inhalation to Subjects With Bronchiolitis
Brief Title: Evaluation of the Safety and Tolerability of Nitric Oxide (NO) Via Inhalation to Subjects With Bronchiolitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beyond Air Inc. (Industry)
Collaborators: Soroka University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AIT_CP_BRONC01.01
Record Dates: First submitted 2013-01-14; First posted 2013-01-16 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-05

CONDITIONS: Bronchiolitis
Keywords: Infants; Bronchiolitis; NO; inhalation
MeSH Terms: conditions — Bronchiolitis; Respiratory Aspiration | interventions — Nitric Oxide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nitric oxide inhalation + standard treatment (Experimental): Inhalation of 160 ppm gNO for 30 minutes, 5 times daily, for 5 consecutive days or until discharged, which occurs first.
  Interventions: Drug: Nitric Oxide
- Standard treatment (Placebo Comparator): Standard treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nitric Oxide
  Arms: Nitric oxide inhalation + standard treatment
Drug: Placebo
  Arms: Standard treatment

SUMMARY:
Prospective, Double Blind, Randomized Single-Center, Evaluation of Safety and Tolerability of Nitric Oxide Given Intermittently via Inhalation to Subjects with Bronchiolitis-Phase IIa Bronchiolitis is defined as an infection of the small airways. It is also the most common manifestation of acute lower respiratory infection (ALRI) in early infancy, and is the leading cause of global child mortality. NO has been shown to play a critical role in various biological functions, including the vasodilatation of smooth muscle, neurotransmission, regulation of wound healing and immune responses to infection such as microbicidal action directed toward various organisms. NO in the airways is considered to play a key role in the innate immune system in which the first-line of host defense against microbes is built.

It has shown the beneficial effect of NO in different diseases with several options of doses and regimens - from newborn with primary pulmonary hypertension which showed improvement in oxygenation after 30 minutes of NO treatment at 10-20 ppm, to a subject with adult respiratory distress syndrome, who demonstrated clinical improvement during NO treatment at 18 and 36 ppm.

In vitro studies utilizing a variety of nitric oxide (NO) donors suggested that NO, in part per million (ppm) concentrations, possesses antimicrobial and anti-viral activity against a wide variety of phyla including bacteria, viruses, helminthes and parasites.

Primary Objectives: Assess the safety of NO intermittent inhalation treatment in 2-12 month old bronchiolitis subjects. Assess the tolerability of NO intermittent inhalation treatment in 2-12 month old bronchiolitis subjects Secondary Objective: Assess the efficacy of NO intermittent inhalation treatment compared to standard treatment in 2-12 months old bronchiolitis subjects.

Prospective, double blind, randomized single-Center study of 44 hospitalized subjects aged 2 -12 months old, diagnosed with bronchiolitis will be enrolled into the study and randomized into 2 groups. Group 1 -Treatment group - Will receive nitric oxide inhalation in addition to standard treatment for up to 5 days, Group 2 - will receive ongoing inhalation of the standard treatment for 5 days.

Treatment administration: Treatment blindness will be kept by separating between unblinded team members (giving the actual treatment) and blinded team members, and by hiding the NO container and all study related equipment behind a curtain. Between study inhalations the subject will continue to receive the standard inhalation treatment. Oxygen (O2), NO , nitrogen dioxide(NO2)and fraction of inspired oxygen (FiO2) delivered to the patient will be continuously monitored.

All subjects will come for follow up visits on day 7(+5), 14 (+5) days and will be contacted on day 30 (+5) from day of admission to the department.

End of study treatment (both groups) will be assessed by a blinded study physician base on clinical assessment. Subject improvement that will lead to end study treatment = clinical score < 6 and/or (Oxygen saturation)SaO2 above 92% and/or decision of subject discharge from the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Subjects (Male or female) 2-12 months old
* Diagnosed as bronchiolitis
* Parents/ legal guardian signed informed consent.

Exclusion Criteria:

* Subjects diagnosed with concomitant diseases such as pneumonia,urine tract infection (UTI) or otitis media
* Prematurity <36 weeks gestational age.
* Received (Respiratory syncytial virus) RSV immunoglobulin prophylaxis
* Subjects diagnosed with, methemoglobinemia, chronic lung disease, immune deficiency, heart disease
* Use of an investigational drug within 30 days before enrollment and not expected to participate in a new study within 30 days
* History of frequent epistaxis (>1 episode/month)
* Significant hemoptysis within 30 days (≥ 5 mL of blood in one coughing episode or > 30 mL of blood in a 24 hour period)
* Methemoglobin >3% at screening
* Subjects cannot fulfill the study design
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the subject or the quality of the data.
* Underlying diseases such as genetic disorders (Cystic fibrosis, Down Syndrome) or chronic lung diseases (Bronchopulmonary dysplasia,Primary ciliary dyskinesia, Bronchiolitis Obliterans), hypotonia, Congenital heart disease)

Ages: 2 Months to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2013-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Met-Hemoglobin percentage (MetHb) associated with inhaled NO | 21 days
Number of participants with adverse events associated with inhaled NO as a measure of safety and tolerability | 5 days

SECONDARY OUTCOMES:
Proportion of subjects (%) who prematurely discontinued the study due to adverse events (AEs) | 5 days

OTHER OUTCOMES:
Comparing the Length of hospital stay (LOS) in days of subjects 2-12 months old with bronchiolitis treated with NO and standard treatment versus subjects treated with standard treatment | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Asher Tal, M.D, Principal Investigator — Soroka University Medical Center
Locations (1):
- Soroka university, Beersheba, Israel